CLINICAL TRIAL: NCT03820596
Title: Safety and Efficacy of Sintilimab(S) in Combination With Histone Deacetylase Inhibitor (Chidamide, C) in Refractory and Relapsed Extranodal Natural Killer Cell/T-cell Lymphoma(EN): A Single-arm, Multicenter Phase I b/II Study(SCENT)
Brief Title: Sintilimab in Combination With Chidamide in Refractory and Relapsed ENKTCL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Huiqiang Huang (Other)
Responsible Party: Sponsor-Investigator, Huiqiang Huang, professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCENT
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Safety and Efficacy
Keywords: Sintilimab; Chidamide; refractory and relapsed; Extranodal natural killer cell/T-cell lymphoma
MeSH Terms: conditions — Recurrence | interventions — sintilimab; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab+Chidamide (Experimental): Sintilimab：200mg(fixed dosage), ivd, qd, q21d
  Chidamide:
  Phase I: 20mg-30mg,biw,continued oral，to evaluate RP2D. Phase II：RP2D，continued oral
  Interventions: Drug: Sintilimab; Drug: Chidamide

INTERVENTIONS:
Drug: Sintilimab — To evaluate the short-term objective efficacy of sintilimab combined with chidamide in the treatment of refractory and relapsed ENKTCL patients, and to determine the MTD, DLT/RP2D of chidamide.
  To evaluate the long-term efficacy and safety of sintilimab combined with chidmide in the treatment of refractory and relapsed ENKTCL patients. Exploring biomarkers that may have predictive effects.
  Other Names: Tyvyt®
Drug: Chidamide — To evaluate the short-term objective efficacy of sintilimab combined with chidamide in the treatment of refractory and relapsed ENKTCL patients, and to determine the MTD, DLT/RP2D of chidamide.
  To evaluate the long-term efficacy and safety of sintilimab combined with chidmide in the treatment of refractory and relapsed ENKTCL patients. Exploring biomarkers that may have predictive effects.
  Other Names: Epidaza

SUMMARY:
Extranodal natural killer/T cell lymphoma(ENKTCL) is a distinct lymphoid neoplasm with aggressive course and poor outcomes. Optimal treatment strategies for advanced ENKTCL have not been fully defined.Patients with disseminated or relapsed disease have a very poor outcome,and there is no standard management for relapsed or refractory disease.Combination chemotherapy remains the mainstay of treatment.In small retrospective studies have observed very good response and survival rates in patients treated with L-asparaginase.In several prospective study that examined relapsed/refractory patients treated with SMILE outside a trial setting,the efficacy sounds good. But treatment related mortality was 7%. The regimen has toxicity, with careful attention to adverse effects and skill acquired through experience. Chidamide, a oral subtype-selective histone deacetylase inhibitor monotherapy was effective on the patients with relapsed or refractory ENKTCL in our study. Objective response rate was 50.0% (6/12) with complete response(CR) rate 33.3 %( 4/12).All four CR patients were still in disease-free more than 6.9 months (6.9-10.5). ENKTCL are invariably infected by Epstein-Barr virus(EBV).EBV-infected lymphoma cells upregulate programmed death ligand 1 (PDL1), ligand of the inhibitory receptor programmed death 1(PD1) on T cells.Ligation of PDL1 on lymphoma cells with PD1 on effector T cells suppresses T-cell cytotoxicity. The PDL1/PD1 axis is therefore a potential mechanism for ENKTCL to avert effector T-cell targeting.PD1 blockadewith pembrolizumab was a potent strategy for ENKTCL failing L-asparaginase regimens in several reports.We carried out a single, open-label, multicenter clinical trial enrolled patients with relapsed or refractory ENKTCL to safety and efficacy of sintilimab in combination With chidamide.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteer to participate in clinical research; fully understand and know the research and sign the Informed Consent Form (ICF); willing to follow and have the ability to complete all trial procedures;
2. Aged 18-75 years old male or female;
3. Extranodal NK/T-cell lymphoma confirmed by histopathology examination;
4. Paraffin tissue specimens or fresh puncture tissue specimens are available;
5. Patients with disease progression or non-remission after asparaginase treatment or asparaginase-contained regimen treatment. Non-remission is defined as: patients did not get partial remission (PR) or better responses after treated by L-asparaginase contained regimen;
6. Eastern cooperative oncology group score: 0-1;
7. Estimated survival ≥ 3 months;
8. There must be at least one evaluate able or measurable lesion that meets the RECIL 2017 Lymphoma criteria [evaluable lesion: 18F-fluorodeoxyglucose/Positron Emission Tomography (18FDG/PET) examination showing increased lymph node or extranodal uptake (higher than liver) and PET and/or computed tomography (Computed Tomography) CT) features are consistent with lymphoma findings; lesions can be measured: nodular lesions > 15mm or extranodal lesions > 10mm (if the only measurable lesion has received radiotherapy in the past, there must be evidence of radiological progress after radiotherapy), and accompanied by increased 18FDG uptake). Except for this, there is no measurable increase in diffuse 18FDG uptake in the liver;
9. Adequate organ and bone marrow function, no severe hematopoietic dysfunction, cardiac, pulmonary, liver, kidney, thyroid dysfunction and immune deficiency (no blood transfusion, granulocyte colony stimulating factor or other medical support was received within 14 days prior to the use of the research drug): 1) The absolute value of neutrophils (>1.0×10^9/L); 2) platelet count (> 75×10^9/L); 3) Hemoglobin (> 9 g/dL); 4) Upper Limit Normal (ULN) or creatinine clearance rate (>40 mL/min) of serum creatinine (<1.5 times normal value upper limit) (estimated by Cockcroft-Gault formula); 5) Serum total bilirubin < 1.5 times ULN; 6) Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT) = 2.5 times ULN; 7) Coagulation function: International Normalized Ratio (INR) = 1.5 times ULN; Prothrombin Time (PT), Activated Partial Thromboplastin Time (APTT) = 1.5 times ULN (unless the subject is receiving anticoagulant therapy and PT and APTT are using anticoagulant therapy at screening time). Within the expected range; 8) Thyrotropin (TSH) or free thyroxine (FT4) or free triiodothyronine (FT3) were all within the normal range (+10%);
10. There was no evidence that subjects had difficulty breathing at rest, and the measured value of pulse oximetry at rest was more than 92%;
11. Participants must pass a pulmonary function test (PFT) to confirm that forced expiratory volume (FEV1)/forced vital capacity (FVC) in the first second is more than 60%, unless it is a large mediastinal mass caused by lymphoma that cannot meet this standard; carbon monoxide diffusion (DLCO), FEV1 and FVC are all above 50% of the predicted value; all PFT results must be obtained within four weeks before the first administration;
12. Subjects who have received antineoplastic therapy should be admitted to the group only after the toxicity of the previous treatment has returned to the level of Common Terminology Criteria for Adverse Events (CTCAE) V5.0 grade score < 1 or baseline level; the level 2 toxicity caused by previous antineoplastic treatment is irreversible and is not expected to deteriorate during the study period. (e.g. thrombocytopenia, anemia, neurotoxicity, alopecia and hearing loss) can be enrolled with the consent of the researchers;
13. Women of Childbearing Potential (WOBCP) must undergo a serum pregnancy test within seven days before the first medication and the results are negative. WOBCP or men and their WOBCP partners should agree to take effective contraceptive measures from the signing of ICF until six months after the last dose of the research drug is used

Exclusion Criteria:

1. Invasive natural killer cell leukemia; 2. Hemophagocytic syndrome; 3. Primary central nervous system lymphoma or secondary central nervous system involvement; 4. Received organ transplantation in the past; 5. Patients who received allogeneic hematopoietic stem cell transplantation within three years before the drug was given (patients who received allogeneic hematopoietic stem cell transplantation more than three years before the drug was given and who currently have no graft-versus-host response can be enrolled); 6. Participating in other clinical studies or planning to start this study is less than 4 weeks from the end of the previous clinical study; 7. Autologous hematopoietic stem cell transplantation was performed within 90 days before the start of the study; 8. The drug was treated with histone deacetylase inhibitors within one year before administration; 9. Patients with active autoimmune diseases requiring systematic treatment in the past two years (hormone replacement therapy is not considered systematic treatment, such as type I diabetes mellitus, hypothyroidism requiring only thyroxine replacement therapy, adrenocortical dysfunction or pituitary dysfunction requiring only physiological doses of glucocorticoid replacement therapy); Patients with autoimmune diseases who do not require systematic treatment within two years can be enrolled; 10. Begin the study on subjects requiring systemic glucocorticoid therapy or other immunosuppressive therapy for a given condition within 14 days before treatment [allowing subjects to use local, ocular, intra-articular, intranasal and inhaled glucocorticoid therapy (with very low systemic absorption); and allowing short-term (< 7 days) glucocorticoid prophylaxis (e.g., contrast agent overdose) Sensitivity) or for the treatment of non-autoimmune diseases (e.g. delayed hypersensitivity caused by contact allergens); 11. In the past five years, patients with other malignant tumors have undergone radical treatment, except for basal cell carcinoma of skin, squamous cell carcinoma of skin, carcinoma in situ of breast and carcinoma in situ of cervix.

12. Begin the study and receive systemic antineoplastic therapy within 28 days before treatment, including chemotherapy, immunotherapy, biotherapy (cancer vaccine, cytokines, or growth factors that control cancer), etc.; 13. The study began with major surgery within 28 days before treatment or radiotherapy within 90 days before treatment; 14. Start the study and receive Chinese herbal medicine or Chinese patent medicine treatment within 7 days before treatment; 15. Begin research on live vaccination (except influenza attenuated vaccine) within 28 days before treatment; 16. History of human immunodeficiency virus (HIV) infection and/or patients with acquired immunodeficiency syndrome are known; 17. Patients with active hepatitis B or active hepatitis C. Patients who are positive for hepatitis B Surface Antigen (HBsAg) or hepatitis C Virus (HCV) antibodies at screening stage must pass further detection of hepatitis B Virus (HBV) DNA titer (no more than 2500 copies/mL or 500 IU/mL) and HCV RNA (no more than the lower limit of the detection method) in the row. In addition to active hepatitis B or hepatitis C infections requiring treatment, group trials can be conducted. Hepatitis B carriers, stable hepatitis B (DNA titer should not be higher than 2500 copies/mL or 500 IU/mL) after drug treatment, and cured hepatitis C patients can be enrolled in the group; 18. Patients with active pulmonary tuberculosis; 19. Start studying any active infections requiring systemic anti-infective treatment within 14 days of treatment.

20. Pregnant or lactating women; 21. People with known history of alcoholism or drug abuse; 22. Have uncontrollable complications, including but not limited to symptomatic congestive heart failure, uncontrollable hypertension, unstable angina, active peptic ulcer or hemorrhagic diseases; 23. History of interstitial lung disease or non-infectious pneumonia. Subjects who had previously had non-infectious pneumonia caused by drugs or radiation but had no symptoms were allowed to enter the group; 24. The QTcF interval is more than 450 msec, unless it is secondary to bundle branch block; 25. Past psychiatric history; incapacitated or restricted; 26. According to the researchers'judgment, patients' underlying condition may increase their risk of receiving research drug treatment, or confuse their judgment on toxic reactions; 27. Other researchers consider it unsuitable for patients to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-29 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Phase 1 Study: Percentage of Participants Experiencing Adverse Events defined as Dose Limiting Toxicities (DLTs) of Chidamide. | Up to 90 days
  Dose-limiting toxicity is defined as protocol-defined chidamide related events within the first 90 days
Phase 1 Study: Maximum tolerable dose of chidamide among participants | Up to 90 days
  Maximum tolerable dose is defined as protocol-defined the highest quantity chidamide among participants.
Phase 1 Study: Maximum tolerable dose(MTD) and recommended Phase 2 dose (RP2D) of chidamide among participants | Up to 90 days
  Maximum tolerable dose is defined as protocol-defined the highest quantity chidamide among participants.
Phase 2 Safety Management Study | Up to12 months
  Incidence and Severity of Toxicities
Efficacy of sintilimab plus chidamide in refractory and relapsed ENKTCL | Up to 24 months
  Objective response including CR and PR rate

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | Up to12 months
  PFS is defined as the time from the treatment date to the date of disease progression per the RECIL 2017 Response Criteria for Malignant Lymphoma or death regardless of cause.
Duration of Response (DOR) | Up to12 months
  Among participants who experience an objective response, DOR is defined as the date of their first objective response (which is subsequently confirmed) to disease progression per the RECIL 2017 Response Criteria for Malignant Lymphoma or Among participants who experience an objective response.
Overall Survival (OS) | Up to 24 months
  OS is defined as the time from treatment to the date of death.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Department of hematology department, Nanfang hospital, Guangzhou, Guangdong
  - Guangdong General Hospital; Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Sun Yat-sen University Cancer Center, Guangzhou